CLINICAL TRIAL: NCT06448286
Title: PH Weighted Chemical Exchange Saturation Transfer Based Surgical Resections of Glioblastoma
Brief Title: PH Weighted Chemical Exchange Saturation Transfer MRI-Based Surgical Resection to Improve Survival in Patients With Glioblastoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-001605; NCI-2024-01961 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy; Contrast Media; Radiotherapy; Radiation; Surgical Procedures, Operative; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, investigators and research staff will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group I (standard of care surgical resection) (Active Comparator): Patients undergo surgical resection with standard intraoperative guidance using contrast-enhanced MRI. Patients also undergo post operative standard of care radiation therapy over 30 fractions and receive standard of care temozolomide PO for 6 weeks. Additionally, patients undergo MRI during follow up.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Procedure: Surgical Procedure; Drug: Temozolomide
- Group II (CEST MRI based surgical resection) (Experimental): Patients undergo surgical resection with intraoperative guidance using CEST MRI. Patients also undergo post operative standard of care radiation therapy over 30 fractions and receive standard of care temozolomide PO for 6 weeks. Additionally, patients undergo MRI during follow up.
  Interventions: Procedure: Chemical Exchange Saturation Transfer Magnetic Resonance Imaging; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Procedure: Surgical Procedure; Drug: Temozolomide

INTERVENTIONS:
Procedure: Chemical Exchange Saturation Transfer Magnetic Resonance Imaging — Undergo CEST MRI
  Other Names: Chemical Exchange Saturation Transfer MRI
  Arms: Group II (CEST MRI based surgical resection)
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo contrast-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI; MRI With Contrast
  Arms: Group I (standard of care surgical resection)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase III trial compares pH weighted chemical exchange saturation transfer (CEST) magnetic resonance imaging (MRI)-based surgical resections to standard of care surgical resections for the treatment of patients with glioblastoma. Standard of care therapy for glioblastoma is surgery to remove tumor tissue that enhances on standard MRI imaging, however, it has been shown that significant tumor burden exists in the region around the tumor tissue that does not enhance with standard MRI. MRI is a procedure in which radio waves and a powerful magnet linked to a computer are used to create detailed pictures of areas inside the body. These pictures can show the difference between normal and tumor tissue. CEST MRI is a technique that uses differences in the tissue environment, like protein concentration or intracellular pH, to generate contrast differences. CEST MRI may identify tumor tissue that does not enhance with standard of care MRI. PH weighted CEST MRI based surgical resection may be more effective compared to standard of care surgical resection in treating patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of potential of hydrogen (pH) sensitive MRI based resections of glioblastoma.

SECONDARY OBJECTIVE:

I. To find surgical and adjuvant therapies to treat infiltrating glioblastoma cells.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo surgical resection with standard intraoperative guidance using contrast-enhanced MRI. Patients also undergo post operative standard of care radiation therapy over 30 fractions and receive standard of care temozolomide orally (PO) for 6 weeks. Additionally, patients undergo MRI during follow up.

GROUP II: Patients undergo surgical resection with intraoperative guidance using CEST MRI. Patients also undergo post operative standard of care radiation therapy over 30 fractions and receive standard of care temozolomide PO for 6 weeks. Additionally, patients undergo MRI during follow up.

After completion of study treatment, patients are followed up at months 3, 6, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Documentation of a newly diagnosed World Health Organization (WHO) grade IV glioblastoma as evidenced by clinical features and imaging data
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Male or female < 18 years of age
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Not medically cleared for surgery
* Previous treatment (any chemotherapy, molecular therapy, immunotherapy, or radiation therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to 2 years
  Multivariate cox and log rank tests will be used to compare progression free survival.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Multivariate cox and log rank tests will be used to compare overall survival.
Surgical complication rate | Up to 2 years
  Independent sample Chi-squared tests will be used to compare differences in surgical complication rate.
Quality of life | Up to 2 years
  Independent sample Chi-squared tests will be used to compare differences in post-operative Karnofsky performance scale changes. The Karnofsky Performance Status (KPS) is a standardized measure used to assess a patient's ability to perform everyday tasks. It ranges from 0 to 100, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Kunal S Patel, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States